CLINICAL TRIAL: NCT02605876
Title: Vibratory Stimuli: A Novel Rehabilitation Method for Preventing Post-traumatic Knee Osteoarthritis
Brief Title: Vibratory Stimuli, A Novel Rehabilitation Method for Preventing Post - Traumatic Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 15-0838
Record Dates: First submitted 2015-11-06; First posted 2015-11-16 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-10

CONDITIONS: Knee Osteoarthritis
Keywords: anterior cruciate ligament reconstruction
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Whole Body Vibration (Experimental): Subjects will receive whole body vibration (30Hz, 2g) applied continuously for 1 minute. This exposure will be repeated 6 times with 2 minutes of rest between exposures.
  Interventions: Device: Whole body vibration
- Local Muscle Vibration (Experimental): Subjects will receive local muscle vibration (30Hz, 2g) applied continuously for 1 minute. This exposure will be repeated 6 times with 2 minutes of rest between exposures.
  Interventions: Device: Local muscle vibration
- Control (No Intervention): Subjects will perform the same procedures as the experimental groups with the exception that no vibratory stimulus will be applied.

INTERVENTIONS:
Device: Whole body vibration
  Arms: Whole Body Vibration
Device: Local muscle vibration
  Arms: Local Muscle Vibration

SUMMARY:
This study will evaluate the acute effects of vibration (whole body vibration and local muscle vibration) on quadriceps function, knee joint proprioception, and gait biomechanics linked to osteoarthritis development in individuals with anterior cruciate ligament reconstruction. Subjects will be randomly assigned to control (no vibration), whole body vibration, and local muscle vibration groups, and the aforementioned characteristics will be assessed prior to and following the respective interventions.

DETAILED DESCRIPTION:
Quadriceps muscle dysfunction and proprioceptive deficits following knee injuries alter walking gait biomechanics in manners that contribute to development of knee osteoarthritis. Current rehabilitation techniques are minimally effective for addressing these complications and preventing knee osteoarthritis. Anterior cruciate ligament reconstruction dramatically increases the risk of knee osteoarthritis, and represents an ideal model for evaluating novel rehabilitation techniques for preventing knee osteoarthritis.

Direct (local muscle vibration) and indirect (whole body vibration) vibratory stimuli enhance quadriceps function and proprioception, and may improve rehabilitation and reduce the risk of knee osteoarthritis. The purpose of this investigation is to determine and compare the acute effects of whole body vibration and local muscle vibration on quadriceps function, knee proprioception, and gait biomechanics in individuals with anterior cruciate ligament reconstruction. The investigators hypothesize that vibratory stimuli will enhance quadriceps function, knee proprioception, and gait biomechanics in manners that would reduce the risk of developing knee osteoarthritis, and that whole body vibration and local muscle vibration will produce equivalent improvements in these characteristics.

ELIGIBILITY:
Inclusion Criteria:

* age 18-35 years
* undergone unilateral ACLR within 5 years prior to participation
* at least 6 months post-ACLR
* Knee Injury and Osteoarthritis Outcome Score (KOOS) self-report survey Pain subscale score > 53.1 and Symptom subscale score > 44.9
* cleared by a physician for return to physical activity, and currently participating in at least 20 minutes of physical activity 3x per week.

Exclusion Criteria:

* central activation ratio (CAR) > 95%
* history of ACL graft rupture or revision surgery, neurological disorder, or injury to either leg within 6 months prior to participation (other than the initial ACLR)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Troy Blackburn, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Neuromuscular Research Lab, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Blackburn T, Padua DA, Pietrosimone B, Schwartz TA, Spang JT, Goodwin JS, Dewig DR, Johnston CD. Vibration improves gait biomechanics linked to posttraumatic knee osteoarthritis following anterior cruciate ligament injury. J Orthop Res. 2021 May;39(5):1113-1122. doi: 10.1002/jor.24821. Epub 2020 Aug 12. PMID 32757272
- [Derived] Blackburn JT, Pietrosimone B, Spang JT, Goodwin JS, Johnston CD. Somatosensory Function Influences Aberrant Gait Biomechanics Following Anterior Cruciate Ligament Reconstruction. J Orthop Res. 2020 Mar;38(3):620-628. doi: 10.1002/jor.24495. Epub 2019 Oct 24. PMID 31608488
- [Derived] Blackburn T, Pietrosimone B, Goodwin JS, Johnston C, Spang JT. Co-activation during gait following anterior cruciate ligament reconstruction. Clin Biomech (Bristol). 2019 Jul;67:153-159. doi: 10.1016/j.clinbiomech.2019.05.010. Epub 2019 May 9. PMID 31121428

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A convenience sample was recruited from local rehabilitation clinics, the University population, the local population, and a nearby Veterans Affairs Medical Center.
Groups:
- Whole Body Vibration: Subjects will receive whole body vibration (30Hz, 2g) applied continuously for 1 minute. This exposure will be repeated 6 times with 2 minutes of rest between exposures.
  Whole body vibration
- Local Muscle Vibration: Subjects will receive local muscle vibration (30Hz, 2g) applied continuously for 1 minute. This exposure will be repeated 6 times with 2 minutes of rest between exposures.
  Local muscle vibration
Period: Overall Study
Arm/Group | Whole Body Vibration | Local Muscle Vibration | Control
Started | 25 | 25 | 25
Completed | 25 | 25 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Whole Body Vibration | Local Muscle Vibration | Control | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 25 | 75
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20 (2) | 20 (3) | 21 (4) | 21 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 17 | 54
  Male | 7 | 6 | 8 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Linear Ground Reaction Force Loading Rate
Description: Change score (Post-Pre) for the ground reaction force during the first 50% of the stance phase calculated as the slope of the vertical ground reaction force time series curve from heelstrike to the first ground reaction force peak. Though a "normal" value has not been established, typical values for the raw scores (i.e. not change scores) range 8.5-9.5 multiples of body weight per second.
Time Frame: Prior to and immediately following vibration interventions (within 5 minutes).
Measure: Mean (95% Confidence Interval); unit: multiples of body weight per second
Arm/Group | Whole Body Vibration | Local Muscle Vibration | Control
Number analyzed (Participants) | 25 | 25 | 25
multiples of body weight per second | 0.276 [0.001 to 0.550] | -0.146 [-0.431 to 0.138] | -0.135 [-0.409 to 0.140]

2. Primary Outcome: Quadriceps Strength
Description: Change score (Post-Pre) for maximal isometric knee extension peak torque in Newton*meters/kilogram body mass. Though a "normal" value has not been established, typical values for the raw values (i.e. not changes scores) range 1.5-3.5 Newton*meters/kilogram body mass.
Time Frame: Prior to and immediately following vibration interventions (within 10 minutes)
Measure: Mean (95% Confidence Interval); unit: Newton*meters/kilogram body mass
Arm/Group | Whole Body Vibration | Local Muscle Vibration | Control
Number analyzed (Participants) | 25 | 25 | 25
Newton*meters/kilogram body mass | 0.05 [-0.04 to 0.15] | -0.13 [-0.23 to -0.03] | -0.09 [-0.19 to 0.01]

3. Primary Outcome: Knee Proprioception
Description: Change score (Post-Pre) for the absolute sagittal plane joint reposition error. This value, measured in degrees, represents the absolute difference between a target knee flexion angle and the angle the subject reproduces, and assesses how well the subject can perceive the position of his/her knee in space. Typical values for the raw scores (i.e. not change scores) range from 0.5 - 5 degrees.
Time Frame: Prior to and immediately following vibration interventions (within 5 minutes)
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Whole Body Vibration | Local Muscle Vibration | Control
Number analyzed (Participants) | 25 | 25 | 25
degrees | -0.71 [-1.15 to -0.27] | -0.61 [-1.06 to -0.16] | -0.08 [-0.53 to 0.38]

4. Primary Outcome: Instantaneous Ground Reaction Force Loading Rate
Description: Change score (Post-Pre) loading rate calculated as the peak of the first time derivative of the vertical ground reaction force time series curve during the first 50% of the stance phase. Though a "normal" value has not been established, typical values for the raw scores (i.e. not change scores) range 50-70 multiples of body weight per second.
Time Frame: Immediately prior to and following the interventions (within 5 minutes)
Measure: Mean (95% Confidence Interval); unit: multiples of body weight per second
Arm/Group | Whole Body Vibration | Local Muscle Vibration | Control
Number analyzed (Participants) | 25 | 25 | 25
multiples of body weight per second | -0.333 [-2.382 to 1.715] | -3.552 [-5.671 to -1.434] | 0.473 [-1.587 to 2.532]

5. Secondary Outcome: Peak Internal Knee Extension Moment
Description: Change score (Post-Pre) for the peak internal knee extension moment during the first 50% of the stance phase. This value reflects the internal (i.e. muscle and other soft tissue) response to external loading of the knee joint in the sagittal plane of motion, and is indicative of quadriceps muscle function during walking. Though a "normal" value has not been established, typical values for the raw scores (i.e. not change scores) range 2-4 % body weight x height.
Time Frame: Immediately prior to and following the interventions (within 5 minutes)
Measure: Mean (95% Confidence Interval); unit: % body weight x height
Arm/Group | Whole Body Vibration | Local Muscle Vibration | Control
Number analyzed (Participants) | 25 | 25 | 25
% body weight x height | 0.271 [0.062 to 0.480] | 0.014 [-0.204 to 0.233] | -0.17 [-0.386 to 0.043]

6. Secondary Outcome: Peak Internal Knee Valgus Moment
Description: Change score (Post-Pre) for the peak internal knee valgus moment during the first 50% of the stance phase. This value reflects the internal (i.e. muscle and other soft tissue) response to external loading of the knee joint in the frontal plane of motion, and is indicative of medial tibiofemoral joint loading during walking. Though a "normal" value has not been established, typical values for the raw scores (i.e. not change scores) range 2-4 % body weight x height.
Time Frame: Immediately prior to and following the interventions (within 5 minutes)
Measure: Mean (95% Confidence Interval); unit: % body weight x height
Arm/Group | Whole Body Vibration | Local Muscle Vibration | Control
Number analyzed (Participants) | 25 | 25 | 25
% body weight x height | -0.450 [-0.750 to -0.061] | -0.436 [-0.795 to -0.077] | -0.304 [-0.660 to 0.051]

ADVERSE EVENTS:
Time Frame: Each participant was enrolled in the study for approximately 3 weeks over which AEs were evaluated. No follow up assessments occurred once participation was complete. Participants were asked to follow up with research team in the event that they experienced any adverse events, but were not directly evaluated.
Arm/Group | Whole Body Vibration | Local Muscle Vibration | Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT02605876/Prot_SAP_000.pdf